CLINICAL TRIAL: NCT01796119
Title: Lateral Alveolar Ridge Expansion in the Maxillary Aesthetic Zone Using Piezo-electric Surgery and Threaded Osteotomes for Immediate Implant Placement.
Brief Title: Ridge Expansion in the Maxillary Aesthetic Zone Using Piezo-electric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Dentaire et d'implantologie Dr.Vinh Nguyen (Other)
Collaborators: Goethe University (Other)
Responsible Party: Principal Investigator, Vinh Giap Nguyen, DDS, D.D.S., Clinique Dentaire et d'implantologie Dr.Vinh Nguyen
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB1665
Record Dates: First submitted 2013-02-18; First posted 2013-02-21 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Tooth Loss
Keywords: Dental implants, Ridge splitting, Ridge expansion
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ridge Splitting (Experimental): Dental implants placed using ridge splitting technique. To measure the horizontal bone width before and after implant insertion and 6 months post-op.
  To measure BLI measured using PA radiographs taken immediately and 6 months post-op.
  To measure implant stability with the resonance frequency analyzer (Osstell,Osstell USA) at time of implant placement, 3 months and 6 months post-op.
  To measure implant success rate. The implants used in this study: NobelActive 3.5 - 4.3mm diameter, 10 - 13 mm in length.
  Interventions: Procedure: Ridge Splitting
- Implants placed using drilling technique (Active Comparator): Dental implants placed in the ridge with sufficient thickness using drilling technique.
  To measure the horizontal bone width before and after implant insertion and 6 months post-op.
  To measure BLI measured using PA radiographs taken immediately and 6 months post-op.
  To measure implant stability with the resonance frequency analyzer (Osstell,Osstell USA) at time of implant placement, 3 months and 6 months post-op.
  To measure implant success rate. The implants used in this study: NobelActive 3.5-4.3mm diameter, 10 - 13 mm in length.
  Interventions: Procedure: Implants placed using drilling technique

INTERVENTIONS:
Procedure: Ridge Splitting — To measure the horizontal bone width before and after implant insertion and 6 months post-op.
  To measure BLI measured using PA radiographs taken immediately and 6 months post-op.
  To measure implant stability with the resonance frequency analyzer (Osstell,Osstell USA) at time of implant placement, 3 months and 6 months post-op.
  To measure implant success rate. The implants used in this study: NobelActive 3.5 - 4.3mm diameter, 10 - 13 mm in length.
  Arms: Ridge Splitting
Procedure: Implants placed using drilling technique — To measure the horizontal bone width before and after implant insertion and 6 months post-op.
  To measure BLI measured using PA radiographs taken immediately and 6 months post-op.
  To measure implant stability with the resonance frequency analyzer (Osstell,Osstell USA) at time of implant placement, 3 months and 6 months post-op.
  To measure implant success rate. The implants used in this study: NobelActive 3.5-4.3mm diameter, 10 - 13 mm in length.
  Arms: Implants placed using drilling technique

SUMMARY:
In this split-mouth controlled study, implants placed using the alveolar ridge expansion technique will be compared to those placed in native bone with sufficient horizontal bone width.

The Piezosurgery device and Bone expanders (Mectron,Italy) will be employed in an alveolar ridge expansion technique.

DETAILED DESCRIPTION:
The success rate of endosseous implant placement in native bone has been proven to be highly predictable. Reliable long term result requires sufficient bone thickness surrounding the implant's body. This is especially true in the maxillary aesthetic zone where buccal bone thickness of 2mm or more is necessary to prevent loss of buccal bone margin and maintain the integrity of the gingival architecture.

Ridge expansion technique, an alternative to bone graft, widens the alveolar ridge prior to implant placement, thus permits the preservation of buccal and lingual bone thickness.

Narrow atrophy edentulous alveolar ridges (study site) in the maxillary aesthetic zone will be split lengthwise using piezo-electric surgery (Piezosurgery, Mectron, USA). The prepared osteotomy will subsequently be expanded using threaded osteotomes (Bone Expanders, Mectron, Italy). Implants will immediately be inserted in the prepared osteotomy. In the edentulous alveolar ridges with sufficient thickness (controlled site) in the maxillary aesthetic zone, implants will be placed directly using conventional drilling technique. Outcome measures will be compared.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Systemically healthy
* Implant therapy will be the elective treatment option.
* The alveolar ridge thickness will be insufficient to receive implant of 3.5-4.3mm in diameter.
* The ridge width will be at least 4mm
* Implants will be placed in the maxillary edentulous ridge from second premolar to the opposite second premolar.
* There will be a second edentulous ridge in the same individual's mouth that serves as control site. The crest of this site will be at least 5.5mm wide, sufficient to receive an implant of 3.5-4.3 mm in diameter.
* Demonstrated ability to maintain oral hygiene
* Willingness and ability to commit to follow-up
* Able to understand study procedure and provide signed informed consent.
* In order to ensure optimal efficacy of the methods used to reduce the risk of pregnancy in female subjects and potential harm to a fetus, contraceptive measures are required in order to participate in the Study, as follows: hormonal methods and the IUD must be in used at least 30 days prior to Study drug administration; that barrier methods must be use in used at least 15 days prior to Study drug administration; that vasectomy must be completed 3 months prior to first Study drug administration; or in the alternative that a 0 sperm count will suffice.

Exclusion Criteria:

* Extreme alveolar ridge atrophy with no cancellous bone between the buccal and palatal cortical plates
* Extensive vertical ridge resorption which requires vertical augmentation
* Uncontrolled periodontal disease.
* Need of sinus lift procedures in the site of intended implant placement.
* Recent febrile illness (within 6 months) that precludes or delays participation
* Wearers of pacemaker.
* Severe renal or liver diseases
* History of radiotherapy of the head and neck region
* Chemotherapy for treatment of malignant tumors at the time of the study.
* Immuno-compromised patients
* Patients on IV bisphosphonates or on long term oral bisphosphonates for more than 3 years.
* Use of disallowed concomitant medications.
* Pregnancy or intending to conceive during the course of the Study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Bucco-lingual bone thickness of the alveolar ridge | 6 months
  To compare the bucco-lingual thickness of the alveolar ridge measured at approximately 1 mm. and 5 mm. below the crestal bone margin, using ridge mapping calipers. These values, measured pre-op, immediately, and 6 months post-op at study site are compared to those measured from controlled site.

SECONDARY OUTCOMES:
To compare BLI measured using PA radiographs | 6 months
  To compare BLI measured using PA radiographs taken immediately, and 6 months post-op at study site. These values are also compared to those measured from controlled site.

OTHER OUTCOMES:
Implant Stability Quotient Values | 3, 6 months
  Implant Stability Quotient Values (Osstell ISQ, Osstell USA) obtained from implants in study site, recording immediately, 3 months and 6 months post-op to evaluate implant stability. These values will also be compared to those obtained from implants placed in controlled site

CONTACTS AND LOCATIONS:
Overall Officials: Vinh Nguyen, DDS., Principal Investigator — Goethe University
Locations (1):
- Clinique Dentaire et d'implantology Dr. Vinh Nguyen, Brossard, Quebec, Canada